CLINICAL TRIAL: NCT04262726
Title: REMOTION: a Randomized Controlled Pilot Trial to Investigate the Feasibility and Potential Effectiveness of a Blended, Transdiagnostic Intervention for Symptom Reduction and Improvement of Emotion Regulation in an Outpatient Psychotherapeutic Setting
Brief Title: REMOTION: a Trial to Investigate the Feasibility and Potential Effectiveness of a Blended, Transdiagnostic Intervention for Symptom Reduction and Improvement of Emotion Regulation in an Outpatient Psychotherapeutic Setting
Acronym: REMOTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-01929
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Mental Disorders
Keywords: Transdiagnostic; Blended therapy; Internet-based; Emotion regulation
MeSH Terms: conditions — Mental Disorders; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REMOTION + TAU (Experimental): Participants in the REMOTION group receive REMOTION in addition to psychotherapy at the outpatient clinic of the Department of Clinical Psychology and Psychotherapy at the University of Bern.
  Interventions: Behavioral: REMOTION; Behavioral: TAU
- TAU (Active Comparator): Participants in TAU receive psychotherapy at the outpatient clinic of the Department of Clinical Psychology and Psychotherapy at the University of Bern.
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: REMOTION — REMOTION is an internet-based intervention aimed at transdiagnostically reducing symptom severity and improving emotion regulation of psychotherapy patients. The structure of REMOTION is based on the idea of an extended process model of emotion regulation as postulated by J.J. Gross (2015). The program includes the following modules: introduction, psychoeducation, identification, selection, implementation and monitoring/modification. A variety of elements based on different psychotherapy approaches (Cognitive Behavioral Therapy, Emotion Focused Therapy, Dialectical Behavior Therapy etc.) are integrated in the program. Participants should work through one module per week. REMOTION is administered as an add-on to treatment as usual (TAU), which is psychotherapy at the outpatient clinic of the Department of Clinical Psychology and Psychotherapy at the University of Bern.
  Arms: REMOTION + TAU
Behavioral: TAU — Treatment as usual (TAU) refers to psychotherapy at the outpatient clinic of the Department of Clinical Psychology and Psychotherapy at the University of Bern. Psychotherapy at the outpatient clinic is based on Psychological Therapy (Grawe, 1998) principles, which are largely rooted in academic psychology and which mainly draw on interventions from Cognitive Behavior Therapy. Individual case conceptualization are key in Psychological Therapy, along with general therapeutic factors and a focus on the therapeutic relationship.

SUMMARY:
Emotion regulation has been identified as an important transdiagnostic factor in the treatment of mental health disorders. This study aims to examine, for the first time, REMOTION, a novel blended therapy intervention aimed at reducing symptom severity and improving emotion regulation of patients in an outpatient psychotherapy setting. REMOTION is an internet based intervention that is administered as an add-on to psychotherapy. This study aims to investigate feasibility and also potential effectiveness of REMOTION in an outpatient setting. Participants will be randomly assigned to the study conditions. Outcomes are assessed at baseline, after six weeks and after twelve weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* In psychotherapeutic treatment at the outpatient clinic of the Department of Clinical Psychology at the University of Bern
* Mental disorder present
* Internet access available
* Written informed consent

Exclusion Criteria:

* Current participation in another intervention, outside of the treatment at the outpatient clinic, that is geared specifically at emotion regulation
* Current or history of psychotic disorders or bipolar disorder
* Acute suicidality
* Insufficient mastery of German language

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2022-11-27 (Actual); Study Completion 2022-11-27 (Actual)

PRIMARY OUTCOMES:
General symptom severity | baseline
  Assessed with Brief Symptom Inventory (Franke, 2000, German version)
General symptom severity | 6 weeks
  Assessed with Brief Symptom Inventory (Franke, 2000, German version)
General symptom severity | 12 weeks
  Assessed with Brief Symptom Inventory (Franke, 2000, German version)

SECONDARY OUTCOMES:
Difficulties in emotion regulation | baseline, 6 weeks,12 weeks
  Assessed with Difficulties in Emotion Regulation Scale (DERS, Gratz & Roemer, 2004, German version by Ehring et al., 2008).
Emotion competencies questionnaire | baseline, 6 weeks, 12 weeks
  Assessed with Emotion Competencies Questionnaire (SEK-27, Berking & Znoj, 2008)
Depressive Symptoms | baseline, 6 weeks, 12 weeks
  Assessed with Patient Health Questionnaire-9 (PHQ-9, German version by Löwe & Spitzer, 2002).
Anxiety symptoms | baseline, 6 weeks, 12 weeks
  Assessed with Generalized Anxiety Disorder Scale-7 (GAD-7, German version by Löwe et al., 2008)
Well-Being | baseline, 6 weeks, 12 weeks
  Assessed with the World Health Organisation-Five Well-Being Index (German version, Brähler, et al., 2007).
Health related quality of life | baseline, 6 weeks, 12 weeks
  Assessed with the Short Form Health Survey (SF-12, German version by Gandek et al., 1998)
Feasibility parameter: number of participants taking part in the study | at randomization
Feasibility parameter: adherence | 6 weeks,12 weeks (REMOTION group only)
  Adherence assessed by amount of modules completed
Feasibility parameter: adherence | 6 weeks,12 weeks (REMOTION group only)
  Adherence assessed by amount of pages visited in REMOTION
Feasibility parameter: adherence | 6 weeks, 12 weeks (REMOTION group only)
  Adherence assessed by amount of exercises completed in REMOTION
Feasibility parameter: program usability | 6 weeks, 12 weeks (REMOTION group only)
  Assessed with the System Usability Scale (SUS, Brooke, 1996)
Feasibility parameter: user experience | 6 weeks, 12 weeks (REMOTION group only)
  Assessed with the meCUE questionnaire (Minge & Riedel, 2013)
Feasibility parameter: attitude toward psychological online interventions | baseline, 6 weeks, 12 weeks
  Attitudes will be assessed with the Attitude toward Psychological Online Interventions Questionnaire (APOI, German version by Schröder, 2015).
Feasibility parameter: satisfaction with the intervention | 6 weeks, 12 weeks (REMOTION group only)
  Assessed with the Client Satisfaction Questionnaire (CSQ-8, German version by Schmidt, 1989, and adapted for internet interventions).

OTHER OUTCOMES:
Therapeutic alliance | 6 weeks, twelve weeks
  Alliance will be assessed with the Working Alliance Inventory (WAI-SR, German version by Wilmers et al., 2008)
Self Compassion | baseline, six weeks, twelve weeks
  Assessed with the Self Compassion Scale (German version by Hupfeld & Ruffieux, 2011)
Negative effects of REMOTION | six weeks, 12 weeks (REMOTION group only)
  Assessed with an adapted version of the Inventory to Assess Negative Effects of Psychotherapy (INEP; Ladwig et al., 2014)
Therapist variables | baseline, 6 weeks, 12 weeks
  Assessed with items created for the study (demographics, use of emotion regulation interventions in therapy, use of online interventions in therapy)
Therapist variables specific to REMOTION | 6 weeks, 12 weeks (REMOTION group only)
  Assessed with items created for the study (for example perceived effect of REMOTION etc.)
Patient emotion regulation difficulties as rated by the therapist | baseline, 6 weeks,12 weeks
  Assessed with the DERS-t (modified version of the German version by Ehring et al., 2008)
Patient emotion regulation competencies as rated by the therapist | baseline, 6 weeks, 12 weeks
  Assessed with the SEK-27-t (modified version of the German version by Bering & Znoj, 2008)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Berger, Prof. Dr., Principal Investigator — Department of Clinical Psychology and Psychotherapy, Institute of Psychology, University of Bern
Locations (1):
- Psychotherapeutische Praxisstelle, Universität Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bielinski LL, Krieger T, Moggi F, Trimpop L, Willutzki U, Nissen C, Berger T. REMOTION Blended Transdiagnostic Intervention for Symptom Reduction and Improvement of Emotion Regulation in an Outpatient Psychotherapeutic Setting: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2020 Nov 12;9(11):e20936. doi: 10.2196/20936. PMID 33180026